CLINICAL TRIAL: NCT02868515
Title: A Clinical Trial to Assess the Effect of Hot Cereal on Digestive Health in Children
Brief Title: The Effect of Hot Cereal on Digestive Health in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PEP-1602
Record Dates: First submitted 2016-06-14; First posted 2016-08-16 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Subjective Measures of Digestive Health Post Consumption
MeSH Terms: interventions — Dietary Fiber

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oatmeal containing beta-glucan (Experimental): 43 g cereal containing 3g fiber per serving
  Interventions: Other: Hot cereal contain 3 g dietary fiber

INTERVENTIONS:
Other: Hot cereal contain 3 g dietary fiber — Intervention involves consumption of a hot cereal over 14 day period

SUMMARY:
The objective of this study is to examine the effects of 2 servings of hot cereal per day over 2 weeks on digestive health in children that typically eat low fiber diets.

DETAILED DESCRIPTION:
Participant eligibility will be screened at visit 1. The study will be a single-arm intervention design. The study procedures will include a pre-study visit, a pre-intervention baseline data collection period, a 14 day intervention period, and an end of study visit.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 7-12 yrs.
* Low fiber eater (<14 g/d)
* Accustomed to eating breakfast at home
* Demonstrates spoken and written English literacy
* Parent/or legal guardian has experience using a cell phone camera
* Parent/or legal guardian is capable of emailing and texting photos by using cell phone features that enable this such as the select and attach option
* Able to provide assent with parent and/or legal guardian after review of study protocol and procedures
* Parent and/or legal guardian will also be required to provide consent on behalf of the child after reviewing study protocol and procedures

Exclusion Criteria:

* Use of enemas, laxatives, proton pump inhibitors, or antibiotics within the past 3 months
* Use of fiber supplements such as fiber gummies (inulin/chicory root), or Metamucil or Citrucel
* Use of vitamin/mineral supplements, multivitamins, or herbal supplements.
* Participation in any other clinical trial up to 6 months before day 1 of participation in this study
* History of medical or surgical events that may significantly affect the study outcomes including diagnosed gastric or digestive diseases
* Not a regular breakfast eater at home
* High-fiber eater (>14 g of fiber per day)
* Allergies to any of the ingredients in the test products
* Children taking medication that affects appetite (i.e. certain ADHD medications that depress appetite)

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-11-15 (Actual); Study Completion 2016-11-15 (Actual)

PRIMARY OUTCOMES:
Self reported frequency scales to questionnaire regarding digestive regularity | 2 weeks

SECONDARY OUTCOMES:
Gastrointestinal tolerance | 2 weeks
  Using questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Slavin, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paruzynski H, Korczak R, Wang Q, Slavin J. A Pilot and Feasibility Study of Oatmeal Consumption in Children to Assess Markers of Bowel Function. J Med Food. 2020 May;23(5):554-559. doi: 10.1089/jmf.2019.0158. Epub 2019 Oct 14. PMID 31613706